CLINICAL TRIAL: NCT02532127
Title: Dentomaxillofacial Paediatric Imaging: An Investigation Towards Low Dose Radiation Induced Risks
Acronym: DIMITRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other); University of Paris 5 - Rene Descartes (Other); Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: S56942
Record Dates: First submitted 2014-12-10; First posted 2015-08-25 (Estimated); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Radiation Dosage
Keywords: Low-dose risk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Saliva sampling (Experimental): Cells will be collected from consenting participants just before and after (30 min and 24 hr) exposure to CBCT, by brushing a swab against the inner cheek, which can be done by the patients themselves. Swab kits are provided together with an envelope for sending the swabs back.
  Interventions: Other: Saliva sampling

INTERVENTIONS:
Other: Saliva sampling — Cells will be collected from consenting participants just before and after (30 min and 24 hr) exposure to CBCT, by brushing a swab against the inner cheek, which can be done by the patients themselves. Swab kits are provided together with an envelope for sending the swabs back.

SUMMARY:
Cone Beam Computed Tomography (CBCT) is an emerging X-ray technology that has found wide applications in dentomaxillofacial imaging. The ability to provide high-resolution 3D images has resulted in a significant increase in the volume of dental radiology procedures. Although CBCT is associated with higher radiation risk to the patient than conventional dental X-ray imaging (intraoral or panoramic), it is considered to be 'low dose' imaging as defined by the High Level Expert Group (HLEG) with doses ranging from a few microsieverts (μSv) to millisieverts (mSv) per examination.

This proposal is set to tackle important issues raised by the HLEG and the Multidisciplinary European Low Dose Initiative (MELODI) platform. In particular, as deduced by the name DIMITRA (Dentomaxillofacial paediatric imaging: an investigation towards low dose radiation induced risks), the project focuses on the uncertainties associated with radiation-induced health risks at low doses in paediatric dentistry and is a multidisciplinary effort to approach the involved risks from different yet interrelated perspectives: radiobiological characterisation, dosimetric quantification, epidemiological surveying and image quality & dose optimization. A unique Monte Carlo simulation (MC) framework will be used to accurately calculate organ doses in dental CBCT imaging, to quantify the radiation induced risk and to feed the radiobiology team with the appropriate data towards the identification, development and validation of biomarkers for radiation induced health effects. Furthermore, it will constitute the basis upon setting up a gender and age related epidemiology study. The balance between image quality and dose levels will be explored aiming at reducing the risk through image quality optimization.

It is expected that DIMITRA's outcomes and deliverables can be presented to a wider forum via a dissemination meeting, leading to further recommendations and potential future adaptations for the use of CBCT in paediatric dentistry.

ELIGIBILITY:
Inclusion Criteria:

* Prospective study with saliva sampling: Patients referred for a CBCT scan from their doctor
* Retrospective study: recorded patients (age 0 - 22) referred to UZ Leuven in the last 2 years including cleft palate patients

Exclusion Criteria:

-

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2014-12; Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Patient-specific dosimetry | dose retrospectively calculated for each patient up to 1 week after irradiation, patients will be followed until the end of the study (May 2017)
  Using a Monte-Carlo based simulator, specifically designed for dental CBCT imaging, adjusted towards specific CBCT geometries and a series of realistic voxel models of paediatric patients will allow the assessment of variability in doses due to differences in anatomy between patients. The organ and effective doses are used for calculating the associated age and gender related cancer risks attributable to dental and maxillofacial CBCT scans.
Saliva sampling | 30 minutes before radiation
Identify and develop biomarkers for radiation-induced health effects | 24 hours after CBCT radiation